CLINICAL TRIAL: NCT06478485
Title: Feasibility and Clinical Applicability of Surgical Segments Choice for Laminoplasty in Multilevel Cervical Spondylotic Myelopathy Guided by Modified K-line and Modified SC-line in MRI
Brief Title: Laminoplasty for Multilevel Cervical Spondylotic Myelopathy Guided by Modified K-line and Modified SC-line in MRI
Status: Recruiting | Type: Observational
Sponsor: Affiliated 2 Hospital of Nantong University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Jiawei Jiang, Department of spine surgery, Affiliated 2 Hospital of Nantong University
Other Study IDs: mK-line and mSC-line
Record Dates: First submitted 2024-06-22; First posted 2024-06-27 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Modified K-line and Modified SC-line in MRI
Keywords: mK-line; mSC-line; Multilevel Cervical Spondylotic Myelopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MCSM: This study collected MRI images and baseline information of patients with multilevel cervical spondylotic myelopathy (MCSM) and underwent Laminoplasty (LAMP) surgery in Nantong First People's Hospital. No interventions would be used. This study just collect the MRI images pre- or postoperation to investigate the effect of the combination of mk-line and mSC-line on the selection of the surgical approach and whether could be used to predict sufficient decompression of cervical spinal cord and clinical outcome in patients after LAMP.
  Interventions: Diagnostic Test: No Intervention: MCSM

INTERVENTIONS:
Diagnostic Test: No Intervention: MCSM — No Intervention: MCSM

SUMMARY:
This study intended to investigate the combined Impact of mK-line and mSC-line on the selection of the surgical approach and whether could be used to predict sufficient decompression of cervical spinal cord and clinical outcome in patients after LAMP.

DETAILED DESCRIPTION:
This study intended to collect MRI of Patients with Multilevel Cervical Spondylotic Myelopathy. K-line(-) patients can be performed LAMP surgery for better prognosis if mK-line(+) and TypeⅠSC-line in MRI, but there are doubts on TypeⅡ and TypeⅢ. However, there has been no study that investigated the combination role of the mK-line and SC-line in surgical decision making for patients with MCSM. In this study, the investigators defined mK-line as a straight line connecting the midpoints of the anteroposterior canal diameter at cranial and caudal vertebrae of the open-door segment in MRI. Accordingly, the investigators propose a modified spinal cord line(mSC-line) that is a straight line connecting the postero-inferior point of the spinal cord at cranial and caudal vertebrae of the open-door segment in MRI, and simplify the mSC-line types into mSC-line(+) and mSC-line(-). In other words, mK-line and mSC-line in MRI are not fixed, but vary depending on the preoperative open-door segments. This study included patients with LAMP surgery for follow up, whose mK-line and mSC-line in MRI were double-positive for preoperative deciding open-door segments.

ELIGIBILITY:
Inclusion Criteria:

(1) Diagnosis of MCSM confirmed by two spine surgeons with MRI examination and clinic signs; (2) More than 2 level lesions and/or spinal stenosis in MRI, underwent LAMP surgery; (3) Available for both preoperative and follow-up imaging data and clinical data, including sex, age, clinical symptoms, Japanese Orthopedic Association (JOA) score, Visual Analog Scale (VAS) score, Neck Disability Index(NDI) score and MRI data.

Exclusion Criteria:

(1) Previous cervical spine surgery; (2) Diagnosis of tumor, central cord syndrome, infection or other acute traumatic injuries; (3) Diagnosed neurological disorders Parkinson's disease, polio, multiple sclerosis, or other central and peripheral nervous system diseases).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators intended to investigate the combined Impact of mK-line and mSC-line on the selection of the surgical approach and whether could be used to predict sufficient decompression of cervical spinal cord and clinical outcome in patients after LAMP.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
sex | From 2020 to 2026
  male or female
age | From 2020 to 2026
  years old, no month or date
Japanese Orthopedic Association (JOA) score | From 2020 to 2026
  The Japanese Orthopaedic Association (JOA) score is widely used to assess the severity of clinical symptoms in patients with cervical compressive myelopathy. Scoring details refer to the Japanese orthopaedic association score (JOA-score modified by Keller 1993)
Visual Analog Scale (VAS) score | From 2020 to 2026
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson.The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. VAS can be presented in a way a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best). Patients points the scores and the investigators recorded.
Neck Disability Index(NDI) score | From 2020 to 2026
  The NDI can be scored as a raw score doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. Points summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage.
  0 points or 0% means : no activity limitations , 50 points or 100% means complete activity limitation.
Cobb angle | From 2020 to 2026
  The Cobb angle is obtained by drawing parallel lines extending from the lower endplate of the most superior vertebral level (C2) and the lower endplate of the most inferior vertebral level (C7).
Ishihara's Cervical Curvature Index(CCI) | From 2020 to 2026
  Ishihara's Cervical Curvature Index(CCI) = (a1 + a2 + a3 + a4)/L*100, where a1 - 4 are the distances between the posterior margins of the inferior endplates of vertebral bodies and a line between the posterior aspects of the inferior endplates of C2 and C7(distance defined as L).

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Cui, Professor, Principal Investigator — Second Affiliated Hospital of Nantong University
Locations (1):
- The Second Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No